CLINICAL TRIAL: NCT06240182
Title: Effect of Piezoelectric Device on Intraoperative Hemorrhage Control and Quality of Life After Endodontic Microsurgery in Maxillary Molar Teeth: a Randomized Controlled Trial
Brief Title: Effect of Piezoelectric Device on Intraoperative Hemorrhage Control and Quality of Life
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Postgraduate Institute of Dental Sciences Rohtak (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Yamini kindra
Record Dates: First submitted 2024-01-15; First posted 2024-02-02 (Actual); Last update posted 2024-02-02 (Actual); Status verified 2024-01

CONDITIONS: Periapical Lesion

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Sham piezoelectric setup for patients undergoing conventional surgery.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Conventional surgery (Active Comparator): performing surgery by surgical carbide burs
  Interventions: Procedure: conventional surgery
- Piezoelectric surgery (Experimental): surgery performed using piezoelectric device
  Interventions: Procedure: piezoelectric device

INTERVENTIONS:
Procedure: conventional surgery — Surgery performed using conventional rotary burs
  Arms: Conventional surgery
Procedure: piezoelectric device — surgery performed using piezoelectric device.
  Arms: Piezoelectric surgery

SUMMARY:
Most osteotomies and apicoectomies in periapical surgeries are performed by surgical carbide or diamond burs. But greater pressure is applied during cutting which causes more thermal and mechanical damage to the bone. Also, when it comes in contact with soft tissues like nerves or vessels it results in profuse bleeding which affects vision in surgery and neurosensory disturbance at a later stage along with the deposition of metal shavings and bony particles resulting in impaired healing. The main advantages of piezoelectric surgery in various studies are highlighted as selective hard tissue cutting and sparing soft tissue, so even if it comes in contact with vessels, nerve or Schneiderian membrane it does not result in profuse bleeding, postoperative nerve damage or perforation.

DETAILED DESCRIPTION:
Most periapical radiolucent lesions heal uneventfully after endodontic treatment. However, some cases may require periradicular surgery in order to remove pathologic tissue from the periapical region and simultaneously eliminate any source of irritation that could not be removed by orthograde root canal treatment

In dentistry, the piezoelectric bone surgery was developed by the oral surgeon Tomaso Vercellotti in 1988, to overcome the limitations of traditional instrumentation, which was first used for maxillary sinus surgery to reduce the incidence of Schneiderian membrane perforations.

Piezoelectric surgery is a promising technical modality with applications in several aspects of endodontic surgery like bone-tissue management, enucleation of radicular cysts, root-end resection & root-end Cavity Preparation. Piezoelectric surgical device operates with principles similar to the piezoelectric dental scaler devices except for its power which is three to six times higher than the piezoelectric dental scalers. The advantages of piezoelectric surgery over conventional endodontic surgery include protection of soft tissues, optimal visualization of the surgical field, decreased blood loss, reduced vibration and noise, increased patient comfort and protection of tooth structures. But some of its disadvantages are initial financial burden for setting up of the unit, long duration of surgery and instruction manuals discouraging its use in patients with cardiac pacemakers.

Less intraoperative blood loss and less chance of inferior alveolar nerve injury was observed on piezoelectric osteotomy in orthognathic surgery at no extra time investment.

In a similar study comparing piezo osteotomy and traditional saw in bimaxillary orthognathic surgery there was significantly reduced blood loss, postoperative hematoma, swelling and nerve impairment in piezo osteotomy but the mean operative time was more

Distance of 1.97mm between the maxillary sinus floor and root apices and even shorter distance between the periapical lesion and maxillary sinus floor warns the surgeon during removal of lesion.

Schneiderian membrane perforation rate while performing lateral window sinus elevation procedure reduced from 30% by conventional surgical burs to 7% by piezoelectric unit.

The capacity of selective cutting, reducing the risk of perforating the sinus lining, and increased visibility of the surgical field due to the cavitation effect from the saline irrigating solution of the piezoelectric unit makes it the preferred option for performing upper molar surgery.

ELIGIBILITY:
Inclusion criteria:

1. Patients between 16-55 years of age
2. ASA-1 or ASA- 2 according to the classification of the American Society of Anesthesiologists)
3. Peri radicular lesion of strictly endodontic origin with size of lesion ≥ 5mm in CBCT
4. non-surgical retreatment unfeasible (post, anatomical complexity, iatrogenic errors) or previously failed treatment.
5. Good periodontal health condition at tooth level.
6. Able to completely understand and sign an informed consent form.

Exclusion criteria:

1. Presence of vertical root fracture
2. Presence of root perforations
3. Miller class III/IV mobility
4. Presence of root resorption
5. Combined endodontic-periodontic lesions.
6. Pregnancy

Ages: 16 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-11-01 (Actual); Primary Completion 2023-04-01 (Actual); Study Completion 2024-05-01 (Estimated)

PRIMARY OUTCOMES:
Quality of life assessment | till 7 days after surgery
  to assess pain, swelling, mouth opening and effect on daily activities of patient among piezosurgery and conventional surgery using patient perception questionnaire
  aon, swelling, mouth opening and any effect on
hemorrhage control | During surgery
  to assess intraoperative hemorrhage control among 2 groups

SECONDARY OUTCOMES:
periapical healing | Base line to 12 months
  periapical healing comparison in 2 groups 2D radiographic healing by Rud et al and Molven et al criteria and 3D healing by modified PENN 3D criteria

CONTACTS AND LOCATIONS:
Overall Officials: DR. Sanjay Tewari, MDS, Study Director — PGIDS,Rohtak, Haryana, 124001
Locations (1):
- PGIDS, Rohtak, Haryana, India